CLINICAL TRIAL: NCT06218589
Title: Non-Invasive Diagnostic Tests for MASLD in Pediatric Population at an Outpatient Clinic: Velacur and Blood-based Novel Tests
Brief Title: Non-Invasive Diagnostic Tests for MASLD in Pediatric Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Sonic Incytes (Industry); The Obesity Society (Other)
Responsible Party: Principal Investigator, Miriam Vos, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00006624
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Metabolic Dysfunction Associated Steatotic Liver Disease; Non-Alcoholic Fatty Liver Disease (NAFLD)
Keywords: Pediatrics
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Velacur Ultrasound (Experimental): Patients 2 to 20 years of age with suspicion of MASLD or presenting to liver clinic for evaluation of liver disease, including possible MASLD receiving a Velacur ultrasound.
  Interventions: Diagnostic Test: Velacur; Diagnostic Test: MRI; Diagnostic Test: Blood sample collection for biomarkers; Diagnostic Test: Liver biopsy

INTERVENTIONS:
Diagnostic Test: Velacur — Velacur is a liver ultrasound that measures hepatic fat and fibrosis through the propagation of a continuously, externally conducted shear wave. An enrolled participant may choose to do the ultrasound at the time of a clinic visit, or research visit or a scheduled radiology visit according to manufacturer's instructions by trained study staff. Fibrosis and steatosis measures will be collected from all scans.
Diagnostic Test: MRI — Participants who have not had an MRI within the past two years will be offered a research MRI (no contrast or sedation will be used) to measure hepatic fat and hepatic stiffness (if required). Participants who have had an MRI or liver biopsy in the past two years will use historical data comparison data. MRI data will include the PDFF hepatic fat, any assessment of fibrosis and notes of other abnormalities.
Diagnostic Test: Blood sample collection for biomarkers — Biomarkers are metabolic thumbprints of how the body is behaving to different health or disease processes, some of the biomarkers can be studied from plasma or serum combined with other demographics. A lipid profile and comprehensive metabolic panel (CMP), if not obtained clinically within 4 weeks, will be collected as a standard of care.
Diagnostic Test: Liver biopsy — Liver biopsy data will be collected only if liver biopsy is done clinically when available and scored using the Nonalcoholic Steatohepatitis Clinical Research Network (NASH CRN) approach.

SUMMARY:
This study aims to test the utility of Velacur ultrasound as a non-invasive, rapid, point of care diagnostic tool for detecting the presence and amount of hepatic steatosis in children and adolescents aged 2 - 20 years.

DETAILED DESCRIPTION:
Non-Alcoholic Fatty Liver Disease (NAFLD) is currently the leading cause of liver disease in children. The name of NAFLD recently changed to metabolic dysfunction associated steatotic liver disease (MASLD). The definition of MASLD is the presence of steatosis in the liver and a metabolic abnormality, in the setting of other liver steatotic liver diseases having been ruled out. Due to its association with obesity and diabetes, MASLD prevalence is rising worldwide following the upward trends of these diseases. Among the United States pediatric population, the prevalence of NAFLD has been measured at around 11% and it varies widely among races. MASLD is likely very similar in numbers. Because of the natural history of the disease, MASLD patients are at risk of developing cardiovascular complications and hepatocellular carcinoma, raising the issue of diagnosing and treating promptly with the most accurate approaches.

Liver biopsy is the gold standard for assessing inflammation and fibrosis in metabolic dysfunction associated steatotic liver disease. This test is highly sensitive and specific, however some weaknesses exist. Liver biopsy uses a small sample size which can misrepresent the overall health/disease of the organ and there can be interpretation variability within the pathologists assessing the histology. Liver biopsy is also an invasive test, making it less desirable due to the potential of complications and cost. Due to these and despite being the most exact test, its invasive nature and its high price, make it not widely used.

There are several clinical needs, including a better way to rapidly diagnose MASLD in the outpatient clinic setting and to measure the severity of MASLD in patients already diagnosed. The first need, to diagnose MASLD requires demonstrating the presence of steatosis through imaging and sending some standard labs to rule out other conditions and assess metabolic features. The second need focuses primarily on fibrosis assessment, because the amount of fibrosis is the most closely associated with long term outcomes. While inflammation quantity is also important for staging MASLD, inflammation tends to rise and fall with changes in lifestyle and presents a less durable finding. Currently, in pediatrics the level of inflammatory injury is reasonably well represented by change in alanine transaminase (ALT). Thus, validating it is not a primary or secondary objective in this proposal.

The most accurate non-invasive imagining diagnostic test for hepatic steatosis in MASLD is Magnetic Resonance Imagining (MRI) and Magnetic Resonance Spectroscopy (MRS). Specifically, the MRI with Proton Density Fat Fraction (PDFF), has shown to have the best results at diagnosing liver steatosis since it is able to map for fat to the whole liver. Accurate fibrosis assessments have been accomplished with the use of Magnetic Resonance Elastography (MRE) and possess an advantage over ultrasound fibrosis measurements because it is independent of abdominal fat. In spite of that, this imaging is not widely available, and it is still highly priced making it less available.

There are a wide variety of ultrasound based tests measuring liver steatosis and it is an inexpensive alternative to diagnose and follow-up patients. Ultrasound is used in conjunction with scores to measure steatosis according to liver echogenicity and visibility of the surrounding organs. Nonetheless, the sensitivity to finding disease decreases for mild cases and only improves when patients have more than 20% hepatocytes that are fatty. Controlled Attenuation Parameter (CAP) in FibroScan machines has been used to address this issue by measuring the ultrasound attenuation and propagation speed of a shear wave delivered by an ultrasound probe (transient elastography, TE). Even though the CAP and TE provide better results, it still has its downfalls in being accurate when the patient is obese and not being extensively accessible.

Velacur is a liver ultrasound that measures hepatic fat and fibrosis through the propagation of a continuously, externally conducted shear wave. Velacur will measure hepatic steatosis and fibrosis through the measures of ultrasound attenuation and the propagation of a shear wave through the liver to measure its stiffness but will perform the stiffness reading using a continuous, externally conducted wave. This technology is thought to provide a better liver volume sample, giving a better reading in obese patients and the software gives live data for easy and fast patient follow-up, making it easy to use from Medical Assistants to Physicians.

There is a need to validate new non-invasive tests to find accurate diagnostic and liver disease staging tools that are simple to use, with easy access and affordable. Due to the small size of the Velacur device and similarity to other technologies available, and the opportunity of collecting blood biomarkers, the investigators want to study the possibility of using both technologies in an outpatient setting to screen and follow up pediatric population with MASLD in Atlanta, Georgia, USA. The investigators will complete a Velacur exam and/or collect blood biomarkers on patients recruited into the study. Statistical analysis will be performed comparing Velacur with the current gold standards of MRI and liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 2-20 years with suspicion of MASLD or presenting to liver clinic for evaluation of liver disease, including possible MASLD
* For participants choosing to do MRI they have to be able to undergo MRI without sedation
* Written/verbal informed consent from parent or legal guardian
* Written/verbal informed assent from the child when indicated by age

Exclusion Criteria:

* Ascites
* Pregnancy
* Failure to give consent or assent
* Have an implanted electronic device such as pacemaker, neurostimulator, or cochlear implant

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Detecting MASLD | Day 1 (day of liver ultrasound)
  The performance of Velacur is assessed as the percentage of correctly identified cases of MASLD (true positives) detected by Velacur imaging. The presence of MASLD will be compared with the determinations from MRI and liver biopsy, the current gold standards.
Specificity of Detecting MASLD | Day 1 (day of liver ultrasound)
  The performance of Velacur is assessed as the percentage of correctly identified lack of MASLD (true negatives) detected by Velacur imaging. The presence of MASLD will be compared with the determinations from MRI and liver biopsy, the current gold standards.
Positive Predictive Value (PPV) | Day 1 (day of liver ultrasound)
  The Positive Predictive Value (PPV) is the ratio of participants who are truly positive for MASLD divided by the number of participants who test positive for MASLD (true positives and false positives).
Negative Predictive Values (NPV) | Day 1 (day of liver ultrasound)
  The Negative Predictive Value (NPV) is the ratio of participants who are truly negative for MASLD divided by the number of participants who test negative for MASLD (true negatives and false negatives).
Area Under the Receiver Operating Curve (ROC) | Day 1 (day of liver ultrasound)
  The area under the receiver operating characteristic curve is used to assess the diagnostic ability of Velacur and MRI in this specific cohort. The area under the ROC ranges from 0 to 1, where 0 indicates that all predictions were incorrect and 1 means that all predictions were correct.
Threshold of Detection Assessed by Youden Index | Day 1 (day of liver ultrasound)
  Thresholds for Velacur to detect MASLD vs non-MASLD (using MRI as the gold standard) will be calculated using the Youden index, maximizing the difference between true positive rate and false positive rate. The Youden Index ranges from 0 to 1 where 1 indicates that there were no false positives or false negatives (the test is perfect) and 0 means that the test is not an effective way to predict the MASLD.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Vos, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Children's Healthcare of Atlanta (CHOA), Atlanta, Georgia
  - Emory Children's Center, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be available for sharing with other researchers including anthropometrics, demographics, laboratory results.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available for sharing after statistical analyses for the main study are complete.
Access Criteria: Researchers interested in using individual participant data from this study should contact the study PI at mvos@emory.edu with a proposal describing how the data will be used. Upon approval of the proposal the data will be sent via secure encrypted email.